CLINICAL TRIAL: NCT07371312
Title: Outcomes of Couples After Failed PGD Management: A Single-Center Study at the Paris PGD Center (Antoine Béclère - Necker)
Acronym: DECOPI
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250912; 2025-A02124-45 (Other: ANSM)
Record Dates: First submitted 2026-01-09; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Infertility
Keywords: Preimplantation Genetic Diagnosis; Assisted Reproductive Technology; Infertility; Reproductive Outcomes; Live Birth; Pregnancy Outcome; Parental Project; Post-treatment Reproductive Pathways; Long-term Outcomes; Couples Reproductive Decisions
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preimplantation genetic testing (PGT) is a reproductive genetic technique aimed at preventing the transmission of severe genetic disorders. In France, its use is strictly regulated and reserved for complex medical situations, often associated with challenging reproductive histories and significant psychological burden.

Despite scientific advances, success rates in preimplantation genetic testing remain limited, making the care pathway a significant source of uncertainty regarding the future of the parental project.

DETAILED DESCRIPTION:
Preimplantation genetic testing (PGT) is a genetic diagnostic procedure performed on one or a few cells biopsied from embryos created through in vitro fertilization (IVF), prior to uterine transfer. The primary aim of PGT is to enable couples at confirmed risk of transmitting a genetic or chromosomal disorder considered to be of particular severity to have a child unaffected by the condition. By offering this possibility, PGT also represents an alternative to prenatal diagnosis (PND) and helps reduce the use of medical termination of pregnancy (MTP) when fetal abnormalities are detected.

In France, PGT is strictly regulated by bioethics laws and the Public Health Code (Article L2131-4). It is authorized only on an exceptional basis, under conditions defined by legislation, for couples at risk of transmitting a serious genetic disorder recognized as incurable at the time of diagnosis (Agence de la biomédecine, 2023). This regulatory framework aims to ensure the ethical and controlled use of this technology. Introduced in France in 1999, PGT is currently performed in only five multidisciplinary centers authorized by the Agence de la biomédecine (ABM): Grenoble, Montpellier, Nantes, Paris, and Strasbourg.

Indications for PGT are diverse and reflect a wide range of medical and familial contexts. They include histories of recurrent pregnancy loss, multiple medical terminations of pregnancy, the presence of a severe genetic disorder in one member of the couple or their offspring, as well as situations in which relatives have been diagnosed with a serious disease or disability, sometimes with late onset. These circumstances are often associated with complex psychological experiences, marked by repeated trauma and high levels of stress. In this context, psychological support is essential throughout the procedure to help couples manage uncertainty and potential treatment failure.

Moreover, despite technological advances, success rates of PGT remain limited. Consequently, the assisted reproductive technology pathway involving PGT represents a major source of stress and may generate significant distress and uncertainty for couples. This process affects individuals on multiple levels: personal, relational, familial, and societal. A better understanding of these factors may allow clinical interventions to be adapted in order to more effectively support couples throughout their care pathway. When the PGT process does not result in the birth of a child, couples are faced with difficult decisions regarding the continuation of their parental project. Several options may then be considered: (i) attempting a natural pregnancy, with or without prenatal diagnosis; (ii) seeking PGT treatment abroad; (iii) considering gamete donation; or (iv) opting for adoption. In some cases, couples choose to discontinue their parental project altogether. Although these trajectories are individual, they are often influenced by medical, social, economic, and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Woman belonging to a couple who initiated at least one ovarian stimulation cycle for IVF (± ICSI) with preimplantation genetic diagnosis (PGD).
* No further PGD-related procedures (oocyte retrieval or embryo transfer) performed in the center after December 31, 2022.
* No live-born child resulting from PGD care.
* Woman who expressed her free and informed non-opposition to participation.

Exclusion Criteria:

* One or more live-born children resulting from PGD care in the center.
* PGD involving gamete donation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women belonging to couples managed for preimplantation genetic diagnosis (PGD) at the Paris PGD center (Hôpital Antoine Béclère - Necker, AP-HP) between 2006 and 2022, whose PGD care was discontinued without resulting in a live birth. Couples are identified from an institutional PGD database. All PGD indications are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of couples with at least one live-born child surviving ≥3 years after failure of preimplantation genetic diagnosis (PGD) | At least 3 years after the failure of PGD care (date of last PGD-related medical procedure in the center)
  Proportion of couples who achieved at least one pregnancy resulting in the birth of a live child who was alive at the age of 3 years or more, following failure of PGD care. PGD failure is defined as the absence of a live-born child resulting from PGD performed in the center. Outcome is assessed based on self-reported data collected via questionnaire, with verification when necessary.

SECONDARY OUTCOMES:
Reason for discontinuation of preimplantation genetic diagnosis (PGD) care | Baseline
  Proportion of couples according to the reason for discontinuation of PGD care (medical decision vs couple's decision), assessed using a self-administered questionnaire.
Continuation of parental project after PGD failure | Baseline
  Proportion of couples who continued or discontinued their parental project after PGD failure, assessed using a self-administered questionnaire.
Post-PGD pathways followed after failure of PGD care | From PGD failure to questionnaire completion
  Description of pathways undertaken after PGD failure, including natural conception attempts, assisted reproductive technology without PGD, PGD in another center, adoption, or abandonment of the parental project, and their outcomes.
Occurrence of at least one pregnancy after PGD failure | From PGD failure to questionnaire completion
  Proportion of couples who achieved at least one pregnancy, whether evolutive or not, after failure of PGD care, regardless of the pathway followed.
Pregnancy occurring at least 3 years after PGD failure | At least 3 years after PGD failure
  Occurrence and date of onset of any pregnancy (evolutive or not) that occurred at least 3 years after the failure of PGD care.
Time to first pregnancy after PGD failure | From PGD failure to date of first pregnancy
  Time interval between the date of the last PGD-related medical procedure performed in the center and the date of onset of the first pregnancy (evolutive or not) obtained after PGD failure.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte SONIGO, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris